CLINICAL TRIAL: NCT06955247
Title: Sensory Motor Integration Versus Bobath Approach on Hand Functions in Hemiplegia Cerebral Palsy Children
Brief Title: Sensory Integration Versus Bobath on Hand Function in Hemiplegia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Radwa Gomaa Abd El aziz Said, physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.RCT/012/005588; radwa gomaa abd el AZIZ (Registry Identifier: radwa gomaa abd el AZIZ)
Record Dates: First submitted 2025-02-27; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Children With Hemiplegia
Keywords: sensory integration; Hand function

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly allocated in to equal two study groups:
  * Study group "1" will receive sensory motor integration in addition to regular physical therapy
  * Study group "2" will receive bobath technique in addition to regular physical therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subjects will be randomly allocated in to equal two study groups: - Study group "1" will receiv (Experimental): Subjects will be randomly allocated in to equal two study groups 26 in each group
  * Study group "1" will receive regular physical therapy for 45 minutes/time in addition to sensory motor integration for 45 minutes/time 3 days per week for 3 months
- - Study group "2" will receive regular physical therapy for 45 minutes/time in addition to bobath (Experimental)
  Interventions: Other: bobath technique

INTERVENTIONS:
Other: sensory motor integration — Study group (1) sensory motor integration for 45 minutes/time ,3 days per week for 3 months Treatment program included two parts; tactile sensation and proprioception stimulation programs. Each of them accounted half of the session and in terms of the type of activity it was divided into three categories: active, passive
Other: bobath technique — *study group ( 2) bobath techniquefor 45 minutes/time 3 days per week for 3 months in the form of:
  1. Preparation phase
  2. Intervention program (Movement facilitation &Functional training)
  Arms: - Study group "2" will receive regular physical therapy for 45 minutes/time in addition to bobath

SUMMARY:
Hand skills do not develop in isolation; it is the result of neurologic development, physiologic maturation and adaptation, and functional development of learned patterns of motion and motor learning Hand skills in HCP are very complex and sensitive as it considered the main issue in playing and achieving milestones, so identification of this problem and its solution is very essential and play a miserable rule in adaptive response which is a basis of child's occupation. so, the current study is conducting to investigate the difference between sensory motor integration approach and bobath technique on hand function as manual dexterity, fine motor precision and fine motor integration on children with hemiplegic cerebral palsy

DETAILED DESCRIPTION:
Sensory integration therapy is the therapeutic mechanism of pediatrics through sensory augmentation which involves the child in enriched playful tasks, promoting a meaningful motor response. The sensory integration theories assume that an affected sensory reception would result in a defect or delay in the development of milestones among children with motor disorders.

The bobath approach provided a new reference aimed to normalize tone and facilitate volitional and automatic movement which tailors based on the patient's individual problems and situational context to manage problems with movement against gravity and postural control Participants will be assigned randomly into two groups of equal number (study group 1 and study group 2 )26 child in each group

* Study group "1" will receive regular physical therapy in addition to sensory motor integration for 45 minutes/time ,3 days per week for 3 months Treatment program included two parts: tactile sensation and proprioception stimulation programs. Each of them accounted half of the session
* Study group"2" will receive regular physical therapy in addition to bobath therapy for 45 minutes/time 3 days per week for 3 months in the form of:

  1. Preparation phase
  2. Intervention program (Movement facilitation &Functional training) base line assessment and after three months re assessment will be taken for both groups using surface electromyography and Bruininks-Oseretsky Test of Motor Proficiency 2nd Edition

ELIGIBILITY:
Inclusion Criteria:

1. Age ranges from 6 to 12 years.
2. Both genders.
3. Diagnosis of hemiplegia.
4. Level II-III on Manual Ability Classification System (MACS)
5. Spasticity grade 2 to 3 on Modified Ashworth Scale (MAS)
6. Level II-III on Gross Motor Classification System (GMCS)

Exclusion Criteria:

1. Significant mental or psychological problems.
2. Significant visual/auditory problem.
3. Botox injection and/or surgery of the affected upper limb in the past 12 months.
4. Surgical procedures of the affected upper limb.
5. Fixed deformities in the affected upper limb.
6. Comorbid physical diseases such as myopathy, neuropathy, and other central and peripheral nervous system disorders.

   -

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Hand functions | 45-60 minutes
  Hand functions as manual dexterity, fine motor precision and fine motor integration will be assessed using Bruininks-Oseretsky Test of Motor Proficiency 2nd Edition

SECONDARY OUTCOMES:
Spasticity | 10 minutes
  Spasticity will be assessed using electromyographic apparatus (H/M ratio )

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy Dokki,Giza Egypt,, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes